CLINICAL TRIAL: NCT02094677
Title: Daily Disposable Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-50
Record Dates: First submitted 2014-03-13; First posted 2014-03-24 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- filcon II 3 and etafilcon A (Active Comparator): Participants were randomized to a test and control lens for each group in a contralateral design.
  Interventions: Device: filcon II 3; Device: etafilcon A
- filcon II 3 and nelfilcon A (Active Comparator): Participants were randomized to a test and control lens for each group in a contralateral design.
  Interventions: Device: filcon II 3; Device: nelfilcon A

INTERVENTIONS:
Device: filcon II 3 — Participants were randomized to wear filcon II 3 test lens.
  Other Names: Hydrogel Daily Disposable Contact Lens
Device: etafilcon A — Participants were randomized to wear etafilcon A control lens.
  Other Names: Hydrogel Daily Disposable Contact Lens; 1 Day Acuvue Moist
  Arms: filcon II 3 and etafilcon A
Device: nelfilcon A — Participants were randomized to wear nelfilcon A control lens.
  Other Names: Hydrogel Daily Disposable Contact Lens; Dailies Aqua Comfort Plus
  Arms: filcon II 3 and nelfilcon A

SUMMARY:
The objective of the study is to compare the overall subjective preference between two Daily Disposable hydrogel lenses when refitted into a third hydrogel lens.

DETAILED DESCRIPTION:
This was a two-day, randomized, non-dispensing, double-masked, contralateral study with two parallel groups. Participants were recruited into one of two groups - participants who habitually wore etafilcon A lens and participants who habitually wore nelfilcon A lens.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual correction and the assigned study lenses;
5. Habitually wears either 1 Day Acuvue Moist or Dailies Aqua Comfort Plus contact lenses.
6. Demonstrates an acceptable fit with the study lenses

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
7. Is aphakic;
8. Has undergone refractive error surgery;

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy four participants were enrolled into the study and 70 participants were randomized and completed the study. 40 were habitual wearers of etafilcon A lens and 30 were habitual wearers of nelfilcon A lens.
Groups:
- Filcon II 3 and Etafilcon A: Participants were randomized to a test and control lens in a contralateral design.
  filcon II 3: Participants were randomized to wear filcon II 3 test lens.
  etafilcon A: Participants were randomized to wear etafilcon A control lens.
- Filcon II 3 and Nelfilcon A: Participants were randomized to a test and control lens in a contralateral design.
  filcon II 3: Participants were randomized to wear filcon II 3 test lens.
  nelfilcon A: Participants were randomized to wear nelfilcon A control lens.
Period: Overall Study
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A
Started | 43 | 31
Completed | 40 | 30
Not Completed | 3 | 1
Not completed — Screening | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (9) | 33.1 (12.4) | 30.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 13 | 7 | 20
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 30 | 70

OUTCOME MEASURES:

1. Primary Outcome: Lens Preference - Filcon II 3 and Etafilcon A or Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens preference of filcon II 3 and etafilcon A or filcon II 3 and nelfilcon A at baseline visit, following insertion, after settling 10-15mins (surveyed at baseline visit) rated by questionnaire.
  (5 possible ratings: Strongly prefer filcon II 3, Slightly prefer filcon II 3, No preference, Slightly prefer etafilcon A/nelfilcon A, Strongly prefer etafilcon A/nelfilcon A).
Time Frame: Baseline visit
Measure: Number; unit: participants
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A
Number analyzed (Participants) | 40 | 30
participants
  Strongly prefer filcon II 3 | 1 | 3
  Slightly prefer filcon II 3 | 14 | 8
  No preference | 8 | 10
  Slightly prefer etafilcon A/nelfilcon A | 8 | 6
  Strongly prefer etafilcon A/nelfilcon A | 9 | 3

2. Primary Outcome: Lens Preference - Filcon II 3 and Etafilcon A or Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens preference of filcon II 3 and etafilcon A after 3 hours lens wear rated by questionnaire. (5 possible ratings: Strongly prefer filcon II 3, Slightly prefer filcon II 3, No preference, Slightly prefer etafilcon A/nelfilcon A, Strongly prefer etafilcon A/nelfilcon A).
Time Frame: 3 hours
Measure: Number; unit: participants
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A
Number analyzed (Participants) | 40 | 30
participants
  Strongly prefer filcon II 3 | 1 | 3
  Slightly prefer filcon II 3 | 10 | 12
  No preference | 7 | 5
  Slightly prefer etafilcon A/nelfilcon A | 13 | 8
  Strongly prefer etafilcon A/nelfilcon A | 9 | 2

3. Primary Outcome: Lens Preference - Filcon II 3 and Etafilcon A or Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens preference of filcon II 3 and etafilcon A after 6 hours lens wear rated by questionnaire (5 possible ratings: Strongly prefer filcon II 3, Slightly prefer filcon II 3, No preference, Slightly prefer etafilcon A/nelfilcon A, Strongly prefer etafilcon A/nelfilcon A).
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A
Number analyzed (Participants) | 40 | 30
participants
  Strongly prefer filcon II 3 | 2 | 5
  Slightly prefer filcon II 3 | 9 | 8
  No preference | 7 | 9
  Slightly prefer etafilcon A/nelfilcon A | 11 | 5
  Strongly prefer etafilcon A/nelfilcon A | 11 | 3

4. Secondary Outcome: Lens Comfort - Filcon II 3 and Etafilcon A
Description: Participant's subjective response for lens comfort of filcon II 3 and etafilcon A after settling 10-15mins (surveyed at baseline visit, 3 hours, and 6 hours) rated by questionnaire (Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever).
Time Frame: Baseline, 3 hours, 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants. Habitual data collected before study lens dispensed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Filcon II 3; Control - Etafilcon A: Participants were randomized to a test and control lens in a contralateral design.
  filcon II 3: Participants were randomized to wear filcon II 3 test lens.
  etafilcon A: Participants were randomized to wear etafilcon A control lens.
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Habitual lens (before study lens dispensed) | 78 (18) | 77 (20)
  Baseline (study lens) | 84 (18) | 90 (10)
  3 hours | 79 (22) | 87 (14)
  6 hours | 75 (24) | 83 (18)

5. Secondary Outcome: Lens Comfort - Filcon II 3 and Nelficon A
Description: Participant's subjective response for lens comfort of filcon II 3 and nelfilcon A after settling 10-15mins (surveyed at baseline visit, 3 hours, and 6 hours) rated by questionnaire (Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever).
Time Frame: Baseline, 3 hours, 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants. Habitual data collected before study lens dispensed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Filcon II 3; Control - Nelfilcon A: Participants were randomized to a test and control lens in a contralateral design.
  filcon II 3: Participants were randomized to wear filcon II 3 test lens.
  nelfilcon A: Participants were randomized to wear nelfilcon A control lens.
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Habitual lens (before study lens dispensed) | 67 (17) | 67 (18)
  Baseline (study lens) | 85 (14) | 88 (14)
  3 hours | 79 (16) | 75 (17)
  6 hours | 76 (24) | 72 (23)

6. Secondary Outcome: Lens Dryness - Filcon II 3 and Etafilcon A
Description: Participant's subjective response for lens dryness of filcon II 3 and etafilcon A (surveyed at 3 and 6 hours after baseline visit) rated by questionnaire (Scale 0-100, 0=cannot be worn, extremely dry 100=no dryness experienced).
Time Frame: 3 hours and 6 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Habitual lens (before study lens dispensed) | 72 (19) | 70 (20)
  3 hours | 78 (24) | 85 (15)
  6 hours | 75 (23) | 82 (18)

7. Secondary Outcome: Lens Dryness - Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens dryness of filcon II 3 and nelfilcon A (surveyed at 3 and 6 hours after baseline visit) rated by questionnaire (Scale 0-100, 0=cannot be worn, extremely dry, 100=no dryness experienced).
Time Frame: 3 hours and 6 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Habitual lens (before study lens dispensedl | 66 (20) | 66 (19)
  3 hours | 79 (16) | 76 (19)
  6 hours | 77 (21) | 74 (23)

8. Secondary Outcome: Lens Handling - Filcon II 3 and Etafilcon A
Description: Participant's subjective response for lens handling of filcon II 3 and etafilcon A following insertion (surveyed at baseline visit) rated by questionnaire (Scale 0-100, 0=very hard to handle causes pain, 100=very easy to handle).
Time Frame: Baseline visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Habitual lens (before study lens dispensed) | 92 (10) | 92 (10)
  Baseline (study lens) | 93 (9) | 91 (10)

9. Secondary Outcome: Lens Handling - Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens handling of filcon II 3 and nelfilcon A following insertion (surveyed at baseline visit) rated by questionnaire (Scale 0-100, 0=very hard to handle, causes pain, 100=very easy to handle).
Time Frame: Baseline visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Habitual lens (before study lens dispensed) | 90 (14) | 90 (14)
  Baseline (study lens) | 92 (14) | 92 (14)

10. Secondary Outcome: Lens Handling (Removal) - Filcon II 3 and Etafilcon A
Description: Participant's subjective response for lens handling of filcon II 3 and etafilcon A following insertion (surveyed 6 hours after baseline visit) rated by questionnaire (Scale 0-100, 0=very hard to handle, causes pain, 100=very easy to handle).
Time Frame: 6 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Habitual lens (before study lens dispensed) | 95 (10) | 95 (10)
  6 hours | 95 (12) | 97 (6)

11. Secondary Outcome: Lens Handling (Removal) - Filcon II 3 and Nelfilcon A
Description: Participant's subjective response for lens handling of filcon II 3 and nelfilcon A following removal (surveyed 6 hours after baseline visit) rated by questionnaire (Scale 0-100, 0=very hard to handle, causes pain, 100=very easy to handle).
Time Frame: 6 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Habitual lens (before study lens dispensed) | 90 (14) | 89 (15)
  6 hours | 94 (16) | 94 (10)

12. Secondary Outcome: Lens Wettability - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens wettability of filcon II 3 and etafilcon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (Scale 0-4, 0.25 increments, 0=excellent wettability, 4=severely reduced wettability).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline | 0.40 (0.73) | 0.33 (0.57)
  6 hours | 0.95 (0.89) | 1.03 (1.12)

13. Secondary Outcome: Lens Wettability - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens wettability of filcon II 3 and nelficon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (Scale 0-4, 0.25 increments, 0=excellent wettability, 4=severely reduced wettability).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.38 (0.46) | 0.25 (0.35)
  6 hours | 0.93 (0.82) | 0.73 (0.79)

14. Secondary Outcome: Lens Fit, Centration - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens fit for centration of filcon II 3 and etafilcon A following insertion (assessed at baseline visit) by biomicroscopy (Optimum or Decentered N T S I).
  N - Nasal, T - Temporal, S - Superior, I - Interior, N/S - Nasal/Superior, N/I - Nasal/Interior, T/S - Temporal/Superior T/I - Temporal/Interior
Time Frame: Baseline
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Number; unit: participants
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
participants
  Optimum | 13 | 13
  N | 0 | 1
  T | 8 | 9
  S | 2 | 4
  I | 5 | 3
  N/S | 0 | 0
  N/I | 0 | 1
  T/S | 5 | 1
  T/I | 7 | 8

15. Secondary Outcome: Lens Fit, Centration - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens fit for centration of filcon II 3 and etafilcon A following insertion (assessed at 6 hours) by biomicroscopy (Optimum or Decentered N T S I) N - Nasal, T - Temporal, S - Superior, I - Interior, N/S - Nasal/Superior, N/I - Nasal/Interior, T/S - Temporal/Superior, T/I - Temporal/Interior
Time Frame: 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Number; unit: participants
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
participants
  Optimum | 16 | 14
  N | 0 | 1
  T | 9 | 9
  S | 2 | 5
  I | 2 | 1
  N/S | 1 | 0
  N/I | 0 | 0
  T/S | 6 | 4
  T/I | 4 | 6

16. Secondary Outcome: Lens Fit, Centration - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens fit for centration of filcon II 3 and nelfilcon A following insertion (assessed at baseline) by biomicroscopy (Optimum or Decentered N T S I) N - Nasal, T - Temporal, S - Superior, I - Interior, N/S - Nasal/Superior, N/I - Nasal/Interior, T/S - Temporal/Superior, T/I - Temporal/Interior
Time Frame: Baseline
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Number; unit: participants
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
participants
  Optimum | 11 | 14
  N | 1 | 0
  T | 3 | 2
  S | 2 | 2
  I | 3 | 2
  N/S | 1 | 1
  N/I | 0 | 2
  T/S | 7 | 4
  T/I | 2 | 3

17. Secondary Outcome: Lens Fit, Centration - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens fit for centration of filcon II 3 and nelfilcon A following insertion (assessed at 6 hours) by biomicroscopy (Optimum or Decentered N T S I) N - Nasal, T - Temporal, S - Superior, I - Interior, N/S - Nasal/Superior, N/I - Nasal/Interior, T/S - Temporal/Superior, T/I - Temporal/Interior
Time Frame: After 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Number; unit: participants
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
participants
  Optimum | 11 | 12
  Nasal | 1 | 1
  T | 4 | 4
  S | 4 | 2
  I | 0 | 1
  N/S | 1 | 1
  N/I | 0 | 1
  T/S | 7 | 4
  T/I | 2 | 4

18. Secondary Outcome: Lens Fit, Post-Blink Movement - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens fit for Post-Blink Movement of filcon II 3 and etafilcon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (measured in Primary Gaze and recorded in 0.1mm steps).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: mm steps
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
mm steps
  Baseline | 0.28 (0.15) | 0.24 (0.15)
  6 hours | 0.30 (0.16) | 0.26 (0.14)

19. Secondary Outcome: Lens Fit, Post-Blink Movement - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens fit for Post-Blink Movement of filcon II 3 and nelfilcon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (measured in Primary Gaze and recorded in 0.1mm steps).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: mm steps
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
mm steps
  Baseline | 0.26 (0.11) | 0.24 (0.10)
  6 hours | 0.23 (0.08) | 0.24 (0.11)

20. Secondary Outcome: Lens Fit, Tightness - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens fit for tightness of filcon II 3 and etafilcon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (Percentage of tightness, 5 increments, 0-100, 0=extremely loose, 100=extremely tight).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: percentage of tightness
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
percentage of tightness
  Baseline | 48 (6) | 50 (6)
  6 hours | 49 (5) | 51 (6)

21. Secondary Outcome: Lens Fit, Tightness - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens fit for tightness of filcon II 3 and nelfilcon A following insertion (assessed at baseline visit and 6 hours) by biomicroscopy (Percentage of tightness, 5 increments, 0-100, 0=extremely loose, 100=extremely tight).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: percentage of tightness
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
percentage of tightness
  Baseline | 50 (7) | 52 (7)
  6 hours | 52 (6) | 53 (8)

22. Secondary Outcome: Lens Surface Deposition - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment for lens surface deposition of filcon II 3 and etafilcon A following insertion (assessed at 6 hour visit) by biomicroscopy (Scale 0-4, 0.25 steps, 0=no deposits, 4=severe deposits).
Time Frame: 6 hour
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale | 0.26 (0.27) | 0.37 (0.47)

23. Secondary Outcome: Lens Surface Deposition - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment for lens surface deposition of filcon II 3 and nelfilcon A following insertion (assessed at 6 hour visit) by biomicroscopy (Scale 0-4, 0.25 steps, 0=no deposits, 4=severe deposits).
Time Frame: 6 hour
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale | 0.27 (0.33) | 0.30 (0.32)

24. Secondary Outcome: High Contrast Visual Acuity - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment of High Contrast Visual Acuity following filcon II 3 and etafilcon A insertion (assessed at baseline visit and 6 hours) by computerized charts. (Positive logMAR values indicate poorer vision, negative values denote better vision than baseline 20/20 value).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
logMAR
  Baseline | -0.08 (0.07) | -0.06 (0.07)
  6 hours | -0.09 (0.07) | -0.07 (0.08)

25. Secondary Outcome: High Contrast Visual Acuity - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment of High Contrast Visual Acuity following filcon II 3 and nelfilcon A insertion (assessed at baseline visit and 6 hours) by computerized charts. (Positive logMAR values indicate poorer vision, negative values denote better vision than baseline 20/20 value)
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Control - Nelilcon A: Participants were randomized to a test and control lens in a contralateral design.
  filcon II 3: Participants were randomized to wear filcon II 3 test lens.
  nelfilcon A: Participants were randomized to wear nelfilcon A control lens.
Arm/Group | Filcon II 3 | Control - Nelilcon A
Number analyzed (Participants) | 30 | 30
logMAR
  Baseline | -0.07 (0.07) | -0.07 (0.07)
  6 hours | -0.08 (0.07) | -0.10 (0.08)

26. Secondary Outcome: Ocular Health, Corneal Staining (Extent) - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment of corneal staining (extent) assessed at screening (before lens insertion) by biomicroscopy (Grade as a % of each zone).
  N - Nasal, T - Temporal, S - Superior, I - Interior, C - Central
Time Frame: 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: percentage of the area of each zone
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
percentage of the area of each zone
  N | 4 (8) | 0 (1)
  T | 1 (6) | 1 (2)
  S | 3 (8) | 2 (5)
  I | 9 (12) | 4 (6)
  C | 0 (2) | 0 (1)

27. Secondary Outcome: Ocular Health, Corneal Staining (Extent) - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment of corneal staining (extent) assessed at 6 hours by biomicroscopy (Grade as a % of each zone).
  N - Nasal, T - Temporal, S - Superior, I - Interior, C - Central
Time Frame: 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: percentage of the area of each zone
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
percentage of the area of each zone
  N | 2 (5) | 2 (5)
  T | 1 (5) | 0 (1)
  S | 2 (5) | 2 (7)
  I | 6 (8) | 4 (5)
  C | 2 (9) | 0 (1)

28. Secondary Outcome: Ocular Health, Conjunctival Hyperemia - Filcon II 3 and Etafilcon A
Description: The ophthalmologist's objective assessment of conjunctival bulbar and limbal hyperemia assessed at screening (before lens insertion) by biomicroscopy (Scale 0-4, 0.5 increments, 0=no redness, 4=redness).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and etafilcon A group which comprises of 40 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Etafilcon A
Number analyzed (Participants) | 40 | 40
units on a scale
  Bulbar | 1.89 (0.38) | 1.81 (0.39)
  Limbal | 1.75 (0.47) | 1.68 (0.51)

29. Secondary Outcome: Ocular Health, Conjunctival Hyperemia - Filcon II 3 and Nelfilcon A
Description: The ophthalmologist's objective assessment of conjunctival bulbar and limbal hyperemia assessed at screening (before lens insertion of filcon II 3 and nelfilcon A) by biomicroscopy (Scale 0-4, 0.5 increments, 0=no redness, 4=redness).
Time Frame: Baseline and 6 hours
Population: These results are between the filcon II 3 and nelfilcon A group which comprises of 30 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon II 3 | Control - Nelfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale
  Bulbar | 1.67 (0.46) | 1.57 (0.29)
  Limbal | 1.35 (0.49) | 1.27 (0.37)

ADVERSE EVENTS:
Time Frame: From dispense up to 2 days for each study lenses
Groups:
- Filcon II 3 and Etafilcon A: Participants wear one of their habitual brand lenses (etafilcon A) in one eye, (comparator) and one comparator lens (filcon II 3) in the other eye.
  filcon II 3: Participants wear one of their habitual brand lenses in one eye (comparator) and one lens of test lens in the other.
  etafilcon A: Participants wear one of their habitual brand lenses in one eye (comparator) and one lens of test lens in the other.
- Filcon II 3 and Nelfilcon A: Participants wear one of their habitual brand lenses (nelfilcon A) in one eye, (comparator) and one comparator lens (filcon II 3) in the other eye.
  filcon II 3: Participants wear one of their habitual brand lenses in one eye (comparator) and one lens of test lens in the other.
  nelfilcon A: Participants wear one of their habitual brand lenses in one eye (comparator) and one lens of test lens in the other.
Arm/Group | Filcon II 3 and Etafilcon A | Filcon II 3 and Nelfilcon A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 0/40 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.